CLINICAL TRIAL: NCT00897832
Title: Developing Predictive Markers of Therapeutic Response in Pancreatic Cancer
Brief Title: Biomarkers in Predicting Response to Treatment in Patients Who Have Undergone Surgery for Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Associate Professor; Radiation Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC GI 0666; P30CA068485 (NIH); VU-VICC-GI-0666; VU-VICC-061225
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pancreatic cancer: Patients with pancreatic cancer
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Using material that is already being acquired as a component of clinical care (only that which is excess after routine clinical care), it will be determined if pre-treatment markers can be used to correlate with clinical outcomes of survival and recurrence. Examples of such markers include studying if the integrity of DNA repair pathway in pancreatic cancers, analyzed by Rad51 and phosphorylated DNA-PK foci formation, correlates with tumor response to radiotherapy, chemotherapy, and overall survival.

SUMMARY:
RATIONALE: Studying samples of tumor tissue in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This laboratory study is looking at biomarkers in predicting response to treatment in patients who have undergone surgery for pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if a method of extracting and identifying biomarkers (i.e., secreted cytokines and growth factors) from tissues of the quantity obtained from typical biopsy can now be applied in the setting of pancreatic cancer
* To correlate pre-treatment biomarkers with recurrence, overall survival, and tumor response to radiotherapy and chemotherapy in patients with pancreatic cancer.

OUTLINE: Tumor tissue specimens are obtained from the Vanderbilt Ingram Cancer Center Human Tissue Acquisition Core and analyzed for biomarkers (e.g., integrity of DNA repair pathways as analyzed by Rad51 and phosphorylated DNA-PK foci formation). The biomarkers are correlated with clinical outcomes (recurrence, overall survival, and tumor response to treatment).

Patients are followed for recurrence, relapse, and death from disease.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of pancreatic cancer
* Excess tissue collected at the time of routine surgery for pancreatic cancer must be available for analysis

Exclusion criteria

* None known

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Determination if a method of extracting and identifying biomarkers from tissues of the quantity obtained from typical biopsy can be applied in the setting of pancreatic cancer | 1 year following final patient data

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee